CLINICAL TRIAL: NCT03134859
Title: Determining Optimal Dosage of Prone Positioning to Facilitate Motor Development and Body Composition in Early Infancy
Brief Title: Determining Optimal Dosage of Prone Positioning in Early Infancy
Acronym: Tummytime
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Erin Wentz PT PhD PCS, Assistant Professor, Department of Physical Therapy, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TTDSUNYMU
Record Dates: First submitted 2017-04-21; First posted 2017-05-01 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Infant Motor Development
Keywords: motor development
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0 to 30 min/day tummy time (Experimental): Group tasked to engage in an accumulation of 0 to 30 minutes of deliberate tummy time activities daily from study entry until the time at which the infant can independently transition in and out of sitting
  Interventions: Behavioral: Tummy Time
- 31-60 min/day tummy time (Experimental): Group tasked to engage in an accumulation of 31 to 60 minutes of deliberate tummy time activities daily from study entry until the time at which the infant can independently transition in and out of sitting
  Interventions: Behavioral: Tummy Time
- >61 min/day tummy time (Experimental): Group tasked to engage in an accumulation of 61 or more minutes of deliberate tummy time activities daily from study entry until the time at which the infant can independently transition in and out of sitting
  Interventions: Behavioral: Tummy Time

INTERVENTIONS:
Behavioral: Tummy Time — deliberate, supervised play time with the baby on his or her front (tummy) when he or she is awake
  Other Names: prone positioning

SUMMARY:
The proposed study is a longitudinal, randomized control trial designed to determine the dosage of daily 'tummy time' needed in early infancy to influence ideal motor development and healthy body composition. Infants will be randomly assigned to one of three 'tummy time' groups: a group prescribed 0 to 30 minutes per day; a group prescribed 31 to 60 minutes per day; and, a group prescribed 61 or more minutes per day. Families will be encouraged to achieve the maximal minutes prescribed for their group and will keep a log of their daily tummy time. Participating infants will be assessed in their home for motor development and body composition at study entry and again every month for 12 months, at 15 months of age and at 18 months of age.

DETAILED DESCRIPTION:
Prone positioning or 'tummy time' in early infancy is advocated as important to support early motor development, improve overall strength, and prevent flattening of the back of the head. The American Academy of Pediatrics state that "a certain amount of prone positioning, or 'tummy time,' while the infant is awake and being observed is recommended to help prevent the development of flattening of the occiput and to facilitate development of the upper shoulder girdle necessary for timely attainment of certain motor milestones." However, specific recommendations on appropriate dosage of prone positioning are not available. In the absence of these specific recommendations, many infants may not be engaging in sufficient 'tummy time' for timely motor development. Moreover, insufficient 'tummy time' is linked to heightened obesity risk in early life. Given the increasing incidence of obesity in infants, primary preventative efforts need to begin early to reduce this risk.

The proposed study is a longitudinal, randomized control trial designed to determine the dosage of daily 'tummy time' needed in early infancy to influence ideal motor development and healthy body composition. Infants will be randomly assigned to one of three 'tummy time' groups: a group prescribed 0 to 30 minutes per day; a group prescribed 31 to 60 minutes per day; and, a group prescribed 61 or more minutes per day. Families will be encouraged to achieve the maximal minutes prescribed for their group and will keep a log of their daily tummy time. Participating infants will be assessed in their home for motor development and body composition at study entry and again every month for 12 months, at 15 months of age and at 18 months of age. Once a participant can independently transition in and out of the sitting position, the family will no longer be responsible for performing deliberate 'tummy time' activities or logging, but monthly motor development and body composition will continue to be monitored until the participant is 18 months of age.

ELIGIBILITY:
Inclusion Criteria:

* full term infants with typical development

Exclusion Criteria:

* premature birth before 37 weeks gestation; known medical condition or diagnosis; any complications that limit full participation in the intervention activities

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Motor Development over time (longitudinal design) | study entry to 18 months of age
  Motor skills as determined by the Bayley Motor Scales, 3rd edition
Ponderal Index over time (longitudinal design) | study entry to 18 months of age
  Estimate of body composition in infants (weight in kg/height in meters cubed)

IPD SHARING:
Plan to Share IPD: No